CLINICAL TRIAL: NCT05962255
Title: The Impact of Slow, Continuous Infusion of Sodium Chloride or Glucose Solution on Diuresis and Urine Composition During Decongestion of Acute Heart Failure Patients
Brief Title: Sodium Chloride vs. Glucose Solute as a Volume Replacement Therapy During Decongestion in Acute Heart Failure
Acronym: SOLVRED-AHF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Gracjan Iwanek, Medical Doctor, Wroclaw Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KB-68/2022
Record Dates: First submitted 2023-06-24; First posted 2023-07-27 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Acute Heart Failure; Congestion; Heart Failure
Keywords: acute heart failure; decongestion; volume replacement; sodium chloride; congestion
MeSH Terms: conditions — Heart Failure | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: 1:1 randomisation to infusion of 0.9% NaCl vs 5% glucose
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.9 % Sodium Chloride solution (Experimental): Patients receiving an intravenous infusion of 0.9% NaCl
  Interventions: Drug: Furosemide intravenous infusion; Drug: Continous intravenous infusion of 0.9% Sodium Chloride solution
- 5% Glucose solution (Active Comparator): Patients receiving an intravenous infusion of 5% glucose
  Interventions: Drug: Furosemide intravenous infusion; Drug: Continous intravenous infusion of 5% Glucose solution

INTERVENTIONS:
Drug: Furosemide intravenous infusion — At baseline, patients will receive a standardised dose of furosemide 1mg/kg (half of the dose administered as bolus and half as in 2h infusion).
  At the 6th and the 12th hour of the study patients will be reassessed and the need for additional diuretics.
Drug: Continous intravenous infusion of 0.9% Sodium Chloride solution — Continuous 48h infusion of 0.9% sodium chloride at a fixed rate v= 83 ml/h x 24h = 2l/24h
  Arms: 0.9 % Sodium Chloride solution
Drug: Continous intravenous infusion of 5% Glucose solution — Continuous 48h infusion of 5% Glucose at a fixed rate v= 83 ml/h x 24h = 2l/24h
  Arms: 5% Glucose solution

SUMMARY:
The aim of the study is to compare the differences in diuretic, natriuretic and clinical response to decongestion in patients receiving different replacement fluid regimens (0.9% sodium chloride vs 5% glucose) in acute heart failure.

ELIGIBILITY:
Inclusion Criteria:

* patients >18 years old who sign the informed consent
* the primary cause of hospitalization is Acute Heart Failure with a need for intravenous Furosemide
* the start of the study within 24h of hospital admission

Exclusion Criteria:

* need for inotropic support
* end stage renal disease on dialysis
* serum sodium > 148mmol/l or < 130 mmol/l.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Urine volume change at individual timepoints during first day of the procedure. | 24 hours
  Comparison of urine volume between the groups at individual timepoints during the first day of the procedure.
Urine volume change at individual timepoints during second day of the procedure. | 48 hours
  Comparison of urine volume between the groups at individual timepoints during the second day of the procedure.
Urine composition at individual time points. | 72 hours
  Comparison of urine composition (urinary sodium and urinary chloride) between the groups and its change during 72h
Cumulative urine output at 24 hours. | 24 hours
  Comparison of cumulative urine output between the groups at 24 hours.
Cumulative urine output at hours. | 48 hours
  Comparison of cumulative urine output between the groups at 48 hours.
Total dose of furosemide. | 48 hours
  Comparison of the total dose of furosemide between the groups at hours.

SECONDARY OUTCOMES:
Total time on intravenous furosemide. | 3 months
  The total time on intravenous furosemide between hospital admission and discharge will be calculated.
Renin-Angiotensin-Aldosterone system activity. | 24 hours
  Comparison of the renin and aldosterone serum levels between the groups at the 24 hours.
Renin-Angiotensin-Aldosterone system activity. | 48 hours
  Comparison of the renin and aldosterone serum levels between the groups at the 48 hours.
Heart Failure rehospitalization | 30 days
  Compare the need for Heart Failure rehospitalization within 30 days.

OTHER OUTCOMES:
Body weight | 24 hours
  Body weight change after the first day of the procedure.
Body weight | 48 hours
  Body weight change after the second day of the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Heart Diseases, Wroclaw Medical University, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biegus J, Iwanek G, Testani J, Zymlinski R, Fudim M, Guzik M, Gajewski P, Ponikowski P. Sodium chloride versus glucose solute as a volume replacement therapy for more effective decongestion in acute heart failure (SOLVRED-AHF): A prospective, randomized, mechanistic study. Eur J Heart Fail. 2025 Nov;27(11):2442-2451. doi: 10.1002/ejhf.3708. Epub 2025 Jun 2. PMID 40455066